CLINICAL TRIAL: NCT04472494
Title: Phase 2, Randomized, Double-Blind Placebo Controlled Study of Intravenous Abatacept in the Treatment of Hospitalized COVID-19 Participants With Respiratory Compromise
Brief Title: Study of Abatacept in the Treatment of Hospitalized COVID-19 Participants With Respiratory Compromise
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-873; U1111-1250-4217 (Other: WHO)
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: Coronavirus disease 2019 (COVID-19); Coronavirus; Coronavirus infections; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abatacept + Standard of care (Experimental)
  Interventions: Biological: Abatacept
- Placebo infusion + Standard of care (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Abatacept — Specified dose on specified days
  Other Names: ORENCIA®; BMS-188667
  Arms: Abatacept + Standard of care
Other: Placebo — Specified dose on specified days
  Arms: Placebo infusion + Standard of care

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intravenous abatacept administered to hospitalized COVID-19 participants with respiratory compromise.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed virological diagnosis of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (by reverse-transcription polymerase chain reaction (RT-PCR)).
* Hospitalized (or in the Emergency Department awaiting a bed after hospitalization)
* Respiratory compromise as defined by requirement of oxygen supplementation to maintain oxygen saturation ≥ 93% but not requiring mechanical ventilation
* Abnormal chest X-ray consistent with COVID-19 and not indicating other serious medical condition that would serve as an exclusionary criteria
* Women and men must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Women who are breastfeeding
* Recent acute infection defined as:

  i) Any acute infection within 60 days prior to randomization that required hospitalization or treatment with parenteral antibiotics (not COVID-19 related) ii) Any acute infection within 30 days prior to randomization that required oral antimicrobial or antiviral therapy
* History of chronic or recurrent bacterial infection (e.g., chronic pyelonephritis, osteomyelitis, bronchiectasis)
* Prior exposure to BMS-188667 (abatacept)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (7):
  - Alternative Research Associates, Llc, Hialeah, Florida
  - Alternative Research Associates, Hialeah, Florida
  - Norton Infectious Disease Institute, Louisville, Kentucky
  - Boston Childrens Hospital, Boston, Massachusetts
  - Local Institution - 0002, Boston, Massachusetts
  - Atlantic Health System, Morristown, New Jersey
  - Methodist Health System Clinical Research Institute (MHSCRI), Dallas, Texas
- Puerto Rico (3):
  - CardioPulmonary Research, Guaynabo
  - Ponce Medical School Foundation, Ponce
  - Fundacion de Investigacion de Diego, San Juan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept: Abatacept 10 mg/kg IV + Standard of care (SOC)
- Placebo: Placebo infusion + Standard of care (SOC)
Period: Pre-treatment
Arm/Group | Abatacept | Placebo
Started (Started = Randomized) | 42 | 19
Completed (Completed = Entering treatment period) | 40 | 19
Not Completed | 2 | 0
Not completed — Other reasons | 2 | 0
Period: Treatment
Arm/Group | Abatacept | Placebo
Started (Started = Entering treatment period) | 40 | 19
Completed (Completed = Completed treatment period) | 34 | 16
Not Completed | 6 | 3
Not completed — Death | 5 | 2
Not completed — Hospital discharge | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 42 | 19 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (14.20) | 60.7 (14.48) | 61.0 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 29 | 13 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 9 | 32
  Not Hispanic or Latino | 19 | 10 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 28 | 10 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Invasive Mechanical Ventilation or Died Prior to or on Day 28
Description: The percentage of participants on invasive mechanical ventilation is defined as the delivery of positive pressure to the lungs via an endotracheal tube (or tracheostomy) or death prior to or on day 28.
Time Frame: From first dose to 28 days post first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Percentage of participants | 30.0 [15.8 to 44.2] | 31.6 [10.7 to 52.5]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.9297, Cochran-Mantel-Haenszel Chi-Square test; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.26 to 4.49]

2. Secondary Outcome: Adjusted Mean Change From Baseline in the Ordinal 8-Point Clinical Status Scale on Day 28
Description: Adjusted mean change from baseline based on the following Ordinal 8-point Clinical Status Scale that was proposed for the National Institute of Allergy and Infectious Diseases (NIAID) Adaptive COVID-19 Treatment Trial (ACTT) and is recorded by the worst score (lowest number) state for each day:
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  3. Hospitalized, on non-invasive mechanical ventilation or high-flow oxygen devices;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  7. Not hospitalized, limitation on activities and/or requiring home oxygen;
  8. Not hospitalized, no limitation on activities Baseline is defined as the last assessment done prior or on Day 1
Time Frame: Baseline and on Day 28
Population: All treated participants
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Score on a scale | 3.20 (0.395) | 2.56 (0.528)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.7400, Cochran-Mantel-Haenszel; Adjusted mean difference from Placebo = 0.64, 95% CI 2-sided [-0.55 to 1.82]

3. Secondary Outcome: Percentage of Participants Who Died
Description: Percentage of participants who died due to any cause. Participants in the following Ordinal 8-point Clinical Status Scale that is recorded by the worst score (lowest number) state for each day meet this definition:
  1) Death
Time Frame: From first dose to 28 days post first dose
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Percentage of participants | 12.5 [2.3 to 22.7] | 15.8 [0.0 to 32.2]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.9684, Cochran-Mantel-Haenszel Chi-Square test; Estimate of Difference = -0.10, 95% CI 2-sided [-20.55 to 20.34] — Estimate of Difference is based on minimum risk weights

4. Secondary Outcome: Percentage of Participants Alive and Free of Respiratory Failure on Day 28±3
Description: Respiratory failure is defined by the type of resources required as defined by the use of any of these: Mechanical ventilation, extracorporeal membrane oxygenation (ECMO) or oxygen delivery by noninvasive positive pressure or high flow nasal cannula.
  Participants in the following Ordinal 8-point Clinical Status Scale that is recorded by the worst score (lowest number) state for each day meet this definition:
  4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitation on activities
Time Frame: Day 28±3
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Percentage of participants | 75.0 [61.6 to 88.4] | 73.7 [53.9 to 93.5]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.8504, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.18 to 3.97]

5. Secondary Outcome: Percentage of Participants Returned to Room Air on Day 28
Description: Recovery of pulmonary function is assessed by the percentage of participants returned to room air on day 28 after they were oxygen dependent and dependence on oxygen has been noted to be prolonged even after hospital discharge.
  Participants in the following Ordinal 8-point Clinical Status Scale that is recorded by the worst score (lowest number) state for each day meet this definition:
  5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 8) Not hospitalized, no limitation on activities
Time Frame: Day 28
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Percentage of participants | 70.0 [55.8 to 84.2] | 57.9 [35.7 to 80.1]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.2724, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.53 to 9.82]
Statistical Analysis 2: Comparison: Abatacept vs Placebo; Test type: Superiority; Estimate of difference = 12.78, 95% CI 2-sided [-10.61 to 36.17]; Estimate of difference is based on minimum risk weights

6. Secondary Outcome: Percentage of Participants Alive and Discharged From the Hospital by Day 28
Description: Percentage of participants alive and discharged from the hospital on day 28. Participants in the following Ordinal 8-point Clinical Status Scale that is recorded by the worst score (lowest number) state for each day meet this definition:
  7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitation on activities
Time Frame: From day 1 up to day 28
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Percentage of participants | 82.5 [70.7 to 94.3] | 73.7 [53.9 to 93.5]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; p = 0.4734, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.33 to 12.64]
Statistical Analysis 2: Comparison: Abatacept vs Placebo; Test type: Superiority; Estimate of difference = 5.43, 95% CI 2-sided [-16.71 to 27.57] — Estimate of difference is based on minimum risk weights

7. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: Percentage of participants with serious adverse events (SAEs). SAE is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life threatening
  * Requires inpatient hospitalization
  * Results in persistent or significant disability
  * Is a congenital anomaly/birth defect
  * Is an important medical event
Time Frame: From first dose to 60 days post first dose
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Percentage of participants | 20.0 | 31.6

8. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) of the Infections and Infestations System Organ Class
Description: Percentage of participants with Serious Adverse Events (SAEs) of the infections and infestations System Organ Class (SOC)
Time Frame: From first dose to 60 days post first dose
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 40 | 19
Percentage of participants | 7.5 | 5.3

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were monitored from first dose to 60 days post last dose (Up to approximately 2 months). Participants were assessed for All Cause Mortality from their date of randomization until the study was completed (up to approximately 11 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Abatacept | Placebo
All-Cause Mortality (participants affected / at risk) | 7/42 | 5/19
Serious Adverse Events (participants affected / at risk) | 8/40 | 6/19
Other Adverse Events (participants affected / at risk) | 8/40 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=40) | Placebo (N=19)
Cardiac arrest (Cardiac disorders) | 3 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Seizure (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=40) | Placebo (N=19)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Mastoid effusion (Ear and labyrinth disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 2
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Urinary tract candidiasis (Infections and infestations) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 1
Troponin I increased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04472494/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT04472494/SAP_001.pdf